CLINICAL TRIAL: NCT05436444
Title: Dose-Escalation Study of a Low Pathogenicity Avian H10N7 Influenza Virus in a Healthy Human Challenge Model
Brief Title: Low Pathogenicity Avian H10N7 Influenza Virus in a Healthy Human Challenge Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 200160; 20-I-0160
Record Dates: First submitted 2022-06-17; First posted 2022-06-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02-20

CONDITIONS: Influenza Infection
Keywords: Influenza A; H10N7; Challenge Model; Influenza; Human Challenge
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): All participants receive challenge virus
  Interventions: Biological: A/Mallard/Ohio-99/MM4/1989 H10N7

INTERVENTIONS:
Biological: A/Mallard/Ohio-99/MM4/1989 H10N7 — The human challenge virus will be administered intranasally to each participant using a nasal atomizer. A total volume of up to 2 mL will be administered split between both nostrils of each participant.

SUMMARY:
Background:

Influenza, also called flu, is a virus. It can cause mild symptoms such as fever, cough, sore throat, and aches. Sometimes, flu can cause serious complications. Researchers want to see how people s immune systems respond to the flu.

Objective:

To find the smallest dose of influenza H10N7 virus that may cause an uncomplicated mild to moderate flu infection in healthy people. This dose will be used in the future to test how well new flu vaccines work.

Eligibility:

Healthy adults age 18-50.

Design:

Participants will be screened with:

Physical exam with vital signs and weight

Medical and medicine review

Blood and urine tests

Electrocardiogram to measure the heart s electrical activity.

Screening tests will be repeated during the study.

Participants will be tested for SARS-CoV-2 and other respiratory infections. For this, a swab will be inserted into the back of the nose.

Participants will be admitted to an isolation room in the Clinical Center. They will stay in the hospital for at least 10 days. They will not have visitors.

Participants may have a heart ultrasound. They may have lung function tests. For this, they will blow into a tube to measure lung capacity.

One dose of the flu virus will be sprayed into participants nostrils. Participants will be monitored 24 hours a day. They will give nasal samples (using nasal washes and brushes) and blood samples almost every day. They will complete surveys about their symptoms.

Participants will be discharged after they have 2 consecutive negative tests for flu.

Participants will have at least 4 follow-up visits: 1 visit every 2 weeks for 8 weeks.

DETAILED DESCRIPTION:
Study Description:

This is a dose-finding and pathogenicity study following human challenge with a low pathogenicity avian influenza A H10N7. Participants will be inoculated with 1 dose of challenge virus during the study and then followed for a minimum of 9 weeks after inoculation. Progressively increasing doses will be used according to a specific plan until either the maximum dose is reached or at least 60% of participants develop mild to moderate influenza disease (MMID).

Objectives:

Primary Objective:

1. Determine the safe dose of A/Mallard/Ohio/99/1989 H10N7 human challenge virus that induces MMID in at least 60% of healthy volunteers or identify the rate of MMID at the maximum dose of 10^7 50% Tissue Culture Infective Dose (TCID50).

Secondary Objective:

1. Evaluate clinical disease, identify clinical markers, and observe initiation of shedding, length of shedding, and pathogenesis in participants with low pathogenicity avian influenza A infection.

Exploratory Objective:

1. Discover viral factors necessary for human infection/adaptation and evaluate host immune response, viral replication, viral fitness, and intrahost evolution.

Endpoints:

Primary Endpoint:

1. Rate of MMID, defined as a positive US Food and Drug Administration (FDA) approved clinical test for influenza plus one or more influenza symptoms.

Secondary Endpoints:

1. Daily and total score on FLU-PRO questionnaire in each participant
2. Number and duration of symptoms and signs elicited by daily oral history and clinical exam
3. Duration and quantity of shedding of influenza in nasal wash/SAM by quantitative real-time polymerase chain reaction (rtPCR).

Exploratory Endpoints:

1. Levels and type of influenza infection induced gene expression determined by human gene expression analysis and high-throughput sequencing.
2. Levels of mucosal and systemic antibodies after inoculation.
3. Change in viral genotype from the inoculum of virus isolated from infected participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

An individual must meet all of the following criteria to be eligible for study participation:

1. Greater than or equal to 18 and less than or equal to 50 years of age.
2. Able to provide consent.
3. Agrees to not use tobacco products, marijuana, or vaping products during participation in this study.
4. Willing to remain in isolation for a minimum of 10 calendar days (or for the duration of viral shedding) and to comply with all study requirements.
5. A male subject is eligible for the study if he meets one of the following criteria, beginning at least 4 weeks prior to enrollment and continuing until 10 weeks after administration of the human challenge virus and follow-up visit #4:

   1. Is infertile, including history of successful vasectomy.
   2. Agrees to practice abstinence.
   3. Agrees that, with heterosexual intercourse with a fertile female partner, he will use a condom with spermicide and his female partner (including those who have undergone bilateral tubal ligation) will use an acceptable form of contraception (see inclusion criterion 6c).
6. A female participant is eligible for this study if she is not pregnant or breastfeeding and meets one of the following criteria, beginning at least 4 weeks prior to enrollment and continuing until 10 weeks after administration of the human challenge virus and follow-up visit #4:

   1. Is infertile, including postmenopausal status (as defined by no menses for greater than or equal to 1 year) or history of hysterectomy.
   2. Agrees to practice abstinence.
   3. Agrees that, with heterosexual intercourse with a fertile male partner, she will use an acceptable form of contraception and her male partner will use a condom with spermicide. Acceptable effective methods of female contraception include the following: bilateral tubal ligation, implant of levonorgestrel, injectable progestogen, intrauterine device, oral contraceptive pills, and diaphragm with spermicide.
7. Willing to have samples stored for future research.
8. Human immunodeficiency virus (HIV) uninfected with a negative test within 60 days of inoculation (Day 0).

EXCLUSION CRITERIA:

An individual meeting any of the following criteria will be excluded from study participation:

1. Has self-reported or medically documented significant medical condition including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression or ongoing malignancy.
   5. Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   6. Post-infectious or post-vaccine neurological sequelae.
2. Has close or household (i.e., share the same apartment or house) high-risk contacts including but not limited to:

   1. Persons greater than or equal to 65 years of age.
   2. Children less than or equal to 5 years of age.
   3. Residents of nursing homes.
   4. Persons of any age with significant chronic medical conditions such as:

      * Chronic pulmonary disease (e.g., asthma).
      * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
      * Chronic medical conditions requiring medical follow-up or hospitalization during the past 5 years (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
      * Immunosuppression or cancer.
      * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
      * Persons who are receiving long-term aspirin therapy.
      * Women who are pregnant, trying to become pregnant, or breastfeeding.
3. Has a body mass index (BMI) less than or equal to 18.5 or greater than or equal to 35.
4. Smokes more than 4 cigarettes or other tobacco products on a weekly basis or any type of vaping/e-cigarette use more than 4 times per week.
5. History of facial reconstructive procedures or nasopharyngeal malformation.
6. Positive for Hepatitis B or Hepatitis C infections.
7. Complete blood count (CBC) with differential outside of the NIH Department of Laboratory Medicine (DLM) normal reference range and deemed clinically significant by the PI.
8. Grade 2 or higher Hemoglobin for female participants or Grade 1 or higher Hemoglobin for male participants.
9. Chemistries in the acute care, mineral, and/or hepatic panels, and/or any of the following: lactate dehydrogenase (LDH), uric acid, creatine kinase, and total protein outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
10. Urinalysis outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
11. Clinically significant abnormality as deemed by the PI on ECG.
12. Clinically significant abnormality as deemed by the PI on ECHO.
13. Clinically significant abnormality as deemed by the PI on the PFT and/or spirometry.
14. Recent acute illness within 1 week of admission to the NIH CC.
15. Known allergy to any component of the interventional agent.
16. Known allergy to treatments for influenza (including but not limited to oseltamivir, nonsteroidals).
17. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
18. Receipt of influenza vaccine within 8 weeks prior to enrollment.
19. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
20. Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
21. Receipt of any unlicensed vaccine within 6 months prior to enrollment.
22. Self-reported or known history of current alcoholism or drug abuse, or positive urine/serum test for drugs of abuse (i.e., amphetamines, cocaine, benzodiazepines, opiates, or metabolites, but not tetrahydrocannabinol or metabolites).
23. Self-reported or known history of psychiatric or psychological issues deemed by the PI to be a contraindication to protocol participation
24. Known close contact with anyone known to have influenza in the past 7 days.
25. Known close contact with anyone known to have COVID-19 in the past 14 days.
26. History of COVID-19-related complications, including, but not limited to: inpatient hospitalization, required the use of oxygen, and/or on-going sequelae.
27. Non-English speaking participants.
28. Any condition that, in the judgment of the PI, is a contraindication to protocol participation or impairs the volunteer s ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
The rate of MMID, defined as a positive FDA-approved clinical test for influenza plus one or more influenza symptoms, is induced. | 9 days
  To determine the dose of A /Mallard/Ohio-99/MM4/1989 H10N7 human challenge virus that induces MMID in at least 60% of healthy volunteers.

SECONDARY OUTCOMES:
Daily and total score on FLUPRO questionnaire and number and duration of symptoms and signs elicited by daily oral history and clinical exam | 28 days
  To evaluate clinical disease, identify clinical markers, and observe initiation of shedding, length of shedding, and pathogenesis in participants

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We are not working with any outside collaborators that require this information.

REFERENCES:
- [Background] Beare AS, Webster RG. Replication of avian influenza viruses in humans. Arch Virol. 1991;119(1-2):37-42. doi: 10.1007/BF01314321. PMID 1863223
- [Background] Memoli MJ, Czajkowski L, Reed S, Athota R, Bristol T, Proudfoot K, Fargis S, Stein M, Dunfee RL, Shaw PA, Davey RT, Taubenberger JK. Validation of the wild-type influenza A human challenge model H1N1pdMIST: an A(H1N1)pdm09 dose-finding investigational new drug study. Clin Infect Dis. 2015 Mar 1;60(5):693-702. doi: 10.1093/cid/ciu924. Epub 2014 Nov 20. PMID 25416753
- [Background] KASEL JA, ALFORD RH, KNIGHT V, WADDELL GH, SIGEL MM. EXPERIMENTAL INFECTION OF HUMAN VOLUNTEERS WITH EQUINE INFLUENZA VIRUS. Nature. 1965 Apr 3;206:41-3. doi: 10.1038/206041a0. No abstract available. PMID 14334358
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0160.html